CLINICAL TRIAL: NCT00534989
Title: Use of FDG PET as Predictor of Residual Disease and Subsequent Relapse in Patients With NHL and HD Undergoing HDC and ASCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr. Naeem A. Chaudhri, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2041-050
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma, Non-Hodgkin; Hodgkin Disease
Keywords: NHL and HD
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease

INTERVENTIONS:
Procedure: FDG PET — FDG PET

SUMMARY:
Cytogenetic Analysis of Bone Marrow Specimen Prior to High Dose Chemotherapy and Autologous Stem Cell Transplantation in Patients with Non-Hodgkin's Lymphoma or Hodgkin's Disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with NHL and HD undergoing HDC and ASCT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Prognosis | overall

CONTACTS AND LOCATIONS:
Overall Officials: Syed Akhtar, MD, Principal Investigator — KFSH & RC